CLINICAL TRIAL: NCT02021279
Title: Evaluation of the Use of Transvaginal Resorbable Biologic Mesh as Compared to Traditional Non-Mesh Surgical Repair for Treating Pelvic Floor Disorders
Brief Title: ACell MatriStem Pelvic Floor Matrix Versus Native Tissue Repair, Comparative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACL2012-001
Record Dates: First submitted 2013-12-20; First posted 2013-12-27 (Estimated); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Pelvic Organ Prolapse
Keywords: pelvic organ prolapse; MatriStem; pelvic floor matrix; ACell; native tissue repair
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MatriStem Pelvic Floor Matrix (Experimental): surgical mesh device
  Interventions: Device: MatriStem Pelvic Floor Matrix
- Native Tissue Repair (Active Comparator): suture repair
  Interventions: Procedure: native tissue repair

INTERVENTIONS:
Device: MatriStem Pelvic Floor Matrix
  Arms: MatriStem Pelvic Floor Matrix
Procedure: native tissue repair
  Other Names: suture repair
  Arms: Native Tissue Repair

SUMMARY:
The primary objective of this study is to assess the safety and effectiveness of MatriStem Pelvic Floor Matrix as compared to native tissue repair for the treatment of pelvic organ prolapse. Patients are evaluated throughout a 3 year follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Subject's leading edge of POP is at or beyond the hymen. At or beyond the hymen is defined as POP-Q scores of Ba ≥ 0 or Bp ≥ 0 or C ≥ 0 (for prolapse of the apical compartment alone) or C ≥ -½ total vaginal length (for a multi-compartment prolapse that includes the apical compartment).
* Subject is seeking surgical intervention for symptomatic POP, which is defined as experiencing symptoms of vaginal bulging or pelvic heaviness. Vaginal bulge or pelvic heaviness will be considered present if a subject responds "yes" (≥1) to PFDI-20, question 3.
* Subject or subject's legally authorized representative is willing to provide written informed consent.
* Subject is willing and able to comply with the follow-up regimen.

Exclusion Criteria:

* Subject has a known hypersensitivity to porcine-based materials (relevant to subjects in MatriStem Pelvic Floor Matrix Group only).
* Subject is pregnant or plans to become pregnant during the study.
* Subject has an active or chronic systemic infection including any gynecologic infection, urinary tract infection (UTI), or tissue necrosis.
* Subject has a known neurologic or medical condition affecting bladder function (e.g. multiple sclerosis, spinal cord injury, or stroke with residual neurologic deficit).
* Subject has chronic systemic pain syndrome (e.g. fibromyalgia, painful bladder syndrome).
* Subject has a systemic connective tissue disease (e.g., scleroderma, systemic lupus erythematous (SLE), Marfans syndrome, Ehlers Danhlos, collagenosis, polymyositis or polymyalgia rheumatica).
* Subject has uncontrolled diabetes mellitus (DM).
* Subject has a history of pelvic organ cancer (e.g. uterine, ovarian, bladder, or cervical).
* Subject has had prior or is currently undergoing radiation, laser therapy, or chemotherapy in the pelvic area.
* Subject has taken systemic steroids (within the last month), immunosuppressive or immunomodulatory treatment (within the last 3 months).
* Subject is seeking obliterative vaginal surgery as treatment for POP (colpoclesis).
* Subject is not able to conform to the modified dorsal lithotomy position.
* Subject is currently participating in or plans to participate in another device or drug study during this study.
* Subject is to planning to undergo concurrent surgical treatment of prolapse using mesh other than the MatriStem Pelvic Floor Matrix.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2014-06-11 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-04-28 (Actual)

PRIMARY OUTCOMES:
The safety and effectiveness of surgical success/failure. | 3 years
  The composite outcome of surgical success evaluates anatomic outcome, patient reported outcome, and no retreatment pelvic organ prolapse.

SECONDARY OUTCOMES:
The surgical success/failure based on an alternate definition of success. | 3 years
  A composite outcome of surgical success based on an alternate definition of anatomic success, patient reported outcome, and no retreatment for pelvic organ prolapse.

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Stanford School of Medicine, Stanford, California
  - Cleveland Clinic FLorida, Weston, Florida
  - Female Pelvic Medicine & Urogynecology, Grand Rapids, Michigan
  - Premier Urology Group, Edison, New Jersey
  - Atlantic Health System, Morristown, New Jersey
  - Princeton Urogynecology, Princeton, New Jersey
  - Garden State Urology, Whippany, New Jersey
  - Premier Medical Group of the Hudson Valley, Poughkeepsie, New York
  - The Christ Hospital, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - The Institute for Female Pelvic Medicine and Reconstructive Surgery, Allentown, Pennsylvania
  - Center for Pelvic Health, Franklin, Tennessee

IPD SHARING:
Plan to Share IPD: No